CLINICAL TRIAL: NCT02641717
Title: Validity of Patient-Collected Wet Mounts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC20150468H
Record Dates: First submitted 2015-12-08; First posted 2015-12-29 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Vaginal Discharge; Trichomonas; Candidiasis; Vaginosis, Bacterial; Vaginitis
Keywords: patient-collected; self-collected; vaginitis; vaginosis, bacterial; candidiasis; trichomonas; vaginal discharge
MeSH Terms: conditions — Vaginal Discharge; Trichomonas Infections; Candidiasis; Vaginosis, Bacterial; Vaginitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): All patients enrolled in this study will self-collect a vaginal swab (experimental) then have a physician collected vaginal swab (gold standard)
  Interventions: Other: vaginal swab

INTERVENTIONS:
Other: vaginal swab

SUMMARY:
Purpose/Objectives: To compare wet mount findings for clue cells, yeast, trichomonads and white blood cells per high-power field in self-collected vaginal specimens, compared to clinician-collected specimens, among symptomatic women visiting the San Antonio Metropolitan Health sexually transmitted disease clinic.

Research Design/Plan: Prospective, non-randomized, non-blinded trial

Methods: Obtain informed consent and specimens from 40 symptomatic adult females (eg abnormal discharge, odor and/or itching). Calculate concordance between clinician- and patient-collected samples using a Wilcoxon Matched-Pair test. Calculate sensitivity, specificity, positive predictive value and negative predictive value of the patient-collected wet mount, using the clinician-collected specimens as the "gold standard."

Clinical Relevance: A "wet mount," or microscopic examination, is commonly used to diagnose trichomoniasis and yeast in females, and constitutes one diagnostic element for bacterial vaginosis. While patient-collected vaginal swabs are acceptable for nucleic acid probe tests for chlamydia and gonorrhea and nucleic acid probe tests for trichomoniasis little information about patient-collected wet mounts exists in the literature. Self-collection by women before being seen by a clinician can increase the speed and efficiency of the visit. The method is highly acceptable to women. In the investigators' clinic, women routinely collect their own gonorrhea and chlamydia swabs, so adding an additional swab would not be burdensome.

DETAILED DESCRIPTION:
Studies have shown that self-collection of vaginal swabs is highly acceptable to women. Studies have also shown that patient-collected vaginal swabs are acceptable for nucleic acid probe tests for chlamydia and gonorrhea and nucleic acid probe tests for trichomoniasis; however, little information about patient-collected wet mounts exists in the literature.

The investigators' goal is to compare wet mount findings for clue cells, yeast, trichomonads and white blood cells per high-power field in self-collected vaginal specimens, compared to clinician-collected specimens, among symptomatic women visiting the San Antonio Metropolitan Health sexually transmitted disease clinic. Self-collection by women before being seen by a clinician can increase the speed and efficiency of the visit. In the investigators' clinic, women routinely collect their own gonorrhea and chlamydia swabs, so adding an additional swab would not be burdensome. Based on the reliability of patient-collected swabs for nucleic amplification tests, it is expected that patient-collected wet mounts could be as valid as conventionally collected samples.

Step-by-Step Methods: Potential study participants as described above will be approached by research staff while in the waiting area. If a patient provides informed consent, she will self-collect a wet mount specimen by inserting a cotton-tip swab in the vagina about 2 inches and rotating for 10-30 seconds; later, her clinician will collect a second specimen from the vaginal fornix and place it in a red-top tube with a small amount of normal saline. The clinician-collected sample will be labeled with the patient's identifying information and processed in the usual way by laboratory staff, with results recorded in electronic medical records. The patient-collected sample will be identified by a number only, and results recorded in a study log. The study is complete when the results of 40 patient- and clinician-collected swabs are recorded.

Data Analysis Plan: Concordance between clinician- and patient-collected samples will be calculated using a Wilcoxon Matched-Pair test. Sensitivity, specificity, positive predictive value and negative predictive value of the patient-collected wet mount will also be calculated, using the clinician-collected specimens as the "gold standard."

ELIGIBILITY:
Inclusion Criteria:

* adult,
* nonpregnant
* females
* with vaginal complaint (ie abnormal discharge, odor, itching)

Exclusion Criteria:

* minors <18 yo
* pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Concordance of patient-collected and clinician-collected wet mounts | to be reviewed immediately at time of collection, documented and specimens discarded. No ongoing comparison, this will only be a single point in time comparison between the physician collected specimen and the patient collected specimen.
  Assess for concordance of clue cells, yeast, trichomonads and white blood cells per high-power field between patient collected vaginal swab and physician collected vaginal swab.

CONTACTS AND LOCATIONS:
Overall Officials: Junda Woo, MD, MPH, Principal Investigator — San Antonio Metropolitan Health District
Locations (1):
- San Antonio Metropolitan Health District, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Workowski KA, Berman S; Centers for Disease Control and Prevention (CDC). Sexually transmitted diseases treatment guidelines, 2010. MMWR Recomm Rep. 2010 Dec 17;59(RR-12):1-110. PMID 21160459
- [Background] Van Der Pol B, Williams JA, Taylor SN, Cammarata CL, Rivers CA, Body BA, Nye M, Fuller D, Schwebke JR, Barnes M, Gaydos CA. Detection of Trichomonas vaginalis DNA by use of self-obtained vaginal swabs with the BD ProbeTec Qx assay on the BD Viper system. J Clin Microbiol. 2014 Mar;52(3):885-9. doi: 10.1128/JCM.02966-13. Epub 2014 Jan 3. PMID 24391200